CLINICAL TRIAL: NCT05403788
Title: Usability Study of a Neuropsychological Intervention Program Based on Virtual Reality in Adults With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporación de Rehabilitación Club de Leones Cruz del Sur (Other)
Collaborators: Colombian School of Engineering Julio Garavito (Other); Universidad del Rosario (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CorporacionRCLCS0007
Record Dates: First submitted 2022-05-27; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; virtual reality; cognitive functions; alpha band; beta band; cerebral lobes; electroencephalography
MeSH Terms: conditions — Parkinson Disease | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with virtual reality (Experimental): Each subject will receive a single session of exercises with the OCULUS QUEST2 (OCULUS VR, USA) and a hand tracking software (Hand Physics Lab, Holonautic, Switzerland). Brain function monitoring will be made by an EEG system ENOBIO 20 (Neuro-electrics, Spain) positioned over subject head. Intervention consisted of exercises with upper limbs and visual feedback. These activities were projected stereoscopically on VR googles.
  Interventions: Device: Intervention with virtual reality

INTERVENTIONS:
Device: Intervention with virtual reality — VR intervention with OCULUS QUEST2 (OCULUS VR, USA) consiste on a VR helmet positioned over subject head. The software consisted of a 3D environment with exercises of upper limbs and visual feedback for the treatment of cognitive and motor dysfunction. The therapist have real-time access to the activities in the 3D environment vby real-time video transmission of the helmet activity.
  The program include a single session. Each session is monitored on safety aspects of the subjects with emphasis on possible side effects of virtual reality.

SUMMARY:
Nowadays, several strategies for treating neuropsychologic function loss in Parkinson disease (PD) have been proposed, such as physical activity performance and developing games to exercise the mind. However, few studies illustrate the incidence of these therapies in neuronal activity. This work aims to study the feasibility of a virtual reality-based program oriented to the cognitive functions' rehabilitation of PD patients. For this, the study was divided in intervention with the program, acquisition of signals, data processing and results analysis.

The study highlights implementing new technologies to rehabilitate people with neurodegenerative diseases.

DETAILED DESCRIPTION:
Nowadays, several strategies for treating neuropsychologic function loss in Parkinson disease (PD) have been proposed, such as physical activity performance and developing games to exercise the mind. However, few studies illustrate the incidence of these therapies in neuronal activity. This work aims to study the feasibility of a virtual reality-based program oriented to the cognitive functions' rehabilitation of PD patients. For this, the study was divided in intervention with the program, acquisition of signals, data processing and results analysis. The alpha and beta bands power behaviour were determined by evaluating the electroencephalography (EEG) signals obtained during the execution of control tests and games of the "Hand Physics Lab" Software, from which five games related to attention, planning, sequencing, concentration, and coordination, were taken.

The study highlights implementing new technologies to rehabilitate people with neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson Disease (Neurologist diagnosed)
* Both gender
* Informed consent accepted
* Adults
* Stage 2 and 3 in the Hoehn Yahr scale

Exclusion Criteria:

* Mental diseases
* Migraines
* Pregnancy

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Power spectral density in the frequency of motor imagery from primary motor cortex | Baseline
  continuous signals will be acquired from the primary motor cortex of lower limbs (FcZ, C2, Cz, C1, Cpz) according to the 10-20 International EEG System. Power spectral density in the frequency band of motor imagery (8-32Hz) will be obtained by OpenVibe Software and Matlab. The measure unit is Decibels per Hertz(dB/Hz).
Power spectral density in the frequency of motor imagery from primary motor cortex Post-Intervention | 2 weeks
  continuous signals will be acquired from the primary motor cortex of lower limbs (FcZ, C2, Cz, C1, Cpz) according to the 10-20 International EEG System. Power spectral density in the frequency band of motor imagery (8-32Hz) will be obtained by OpenVibe Software and Matlab. The measure unit is Decibels per Hertz(dB/Hz).

CONTACTS AND LOCATIONS:
Overall Officials: Patricio E Barría Aburto, MSc., Principal Investigator — Corporación de Rehabilitacion Club de Leones Cruz del Sur
Locations (1):
- Corporación de Rehabilitación Club de Leones Cruz del Sur, Punta Arenas, Region of Magallanes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tysnes OB, Storstein A. Epidemiology of Parkinson's disease. J Neural Transm (Vienna). 2017 Aug;124(8):901-905. doi: 10.1007/s00702-017-1686-y. Epub 2017 Feb 1. PMID 28150045
- [Background] Sveinbjornsdottir S. The clinical symptoms of Parkinson's disease. J Neurochem. 2016 Oct;139 Suppl 1:318-324. doi: 10.1111/jnc.13691. Epub 2016 Jul 11. PMID 27401947
- [Background] Hirsch L, Jette N, Frolkis A, Steeves T, Pringsheim T. The Incidence of Parkinson's Disease: A Systematic Review and Meta-Analysis. Neuroepidemiology. 2016;46(4):292-300. doi: 10.1159/000445751. Epub 2016 Apr 23. PMID 27105081
- [Background] Navaratnam P, Arcona S, Friedman HS, Leoni M, Shaik S, Sasane R. Natural history and patterns of treatment change in Parkinson's disease: A retrospective chart review. Clin Park Relat Disord. 2021 Dec 8;6:100125. doi: 10.1016/j.prdoa.2021.100125. eCollection 2022. PMID 34950865
- [Background] Tran TN, Ha UNL, Nguyen TM, Nguyen TD, Vo KNC, Dang TH, Trinh PMP, Truong D. The effect of Non-Motor symptoms on Health-Related quality of life in patients with young onset Parkinson's Disease: A single center Vietnamese Cross-Sectional study. Clin Park Relat Disord. 2021 Nov 24;5:100118. doi: 10.1016/j.prdoa.2021.100118. eCollection 2021. PMID 34927047
- [Background] Weintraub D, Claassen DO. Impulse Control and Related Disorders in Parkinson's Disease. Int Rev Neurobiol. 2017;133:679-717. doi: 10.1016/bs.irn.2017.04.006. Epub 2017 Jun 1. PMID 28802938
- [Background] Duchesne C, Lungu O, Nadeau A, Robillard ME, Bore A, Bobeuf F, Lafontaine AL, Gheysen F, Bherer L, Doyon J. Enhancing both motor and cognitive functioning in Parkinson's disease: Aerobic exercise as a rehabilitative intervention. Brain Cogn. 2015 Oct;99:68-77. doi: 10.1016/j.bandc.2015.07.005. Epub 2015 Aug 7. PMID 26263381
- [Background] Wen D, Lan X, Zhou Y, Li G, Hsu SH, Jung TP. The Study of Evaluation and Rehabilitation of Patients With Different Cognitive Impairment Phases Based on Virtual Reality and EEG. Front Aging Neurosci. 2018 Apr 3;10:88. doi: 10.3389/fnagi.2018.00088. eCollection 2018. No abstract available. PMID 29666577
- [Background] Cikajlo I, Peterlin Potisk K. Advantages of using 3D virtual reality based training in persons with Parkinson's disease: a parallel study. J Neuroeng Rehabil. 2019 Oct 17;16(1):119. doi: 10.1186/s12984-019-0601-1. PMID 31623622
- [Background] Alarcon G, Guy CN, Binnie CD. A simple algorithm for a digital three-pole Butterworth filter of arbitrary cut-off frequency: application to digital electroencephalography. J Neurosci Methods. 2000 Dec 15;104(1):35-44. doi: 10.1016/s0165-0270(00)00324-1. PMID 11163409
- [Background] Zietsch BP, Hansen JL, Hansell NK, Geffen GM, Martin NG, Wright MJ. Common and specific genetic influences on EEG power bands delta, theta, alpha, and beta. Biol Psychol. 2007 May;75(2):154-64. doi: 10.1016/j.biopsycho.2007.01.004. Epub 2007 Jan 25. PMID 17316957
- [Background] Armstrong RA. Visual symptoms in Parkinson's disease. Parkinsons Dis. 2011;2011:908306. doi: 10.4061/2011/908306. Epub 2011 May 25. PMID 21687773
- [Background] Bronte-Stewart H, Barberini C, Koop MM, Hill BC, Henderson JM, Wingeier B. The STN beta-band profile in Parkinson's disease is stationary and shows prolonged attenuation after deep brain stimulation. Exp Neurol. 2009 Jan;215(1):20-8. doi: 10.1016/j.expneurol.2008.09.008. Epub 2008 Sep 27. PMID 18929561
- [Background] Botha H, Carr J. Attention and visual dysfunction in Parkinson's disease. Parkinsonism Relat Disord. 2012 Jul;18(6):742-7. doi: 10.1016/j.parkreldis.2012.03.004. Epub 2012 Apr 11. PMID 22503538
- [Background] Magosso E, De Crescenzio F, Ricci G, Piastra S, Ursino M. EEG Alpha Power Is Modulated by Attentional Changes during Cognitive Tasks and Virtual Reality Immersion. Comput Intell Neurosci. 2019 Jun 25;2019:7051079. doi: 10.1155/2019/7051079. eCollection 2019. PMID 31341468
- [Background] Gola M, Magnuski M, Szumska I, Wrobel A. EEG beta band activity is related to attention and attentional deficits in the visual performance of elderly subjects. Int J Psychophysiol. 2013 Sep;89(3):334-41. doi: 10.1016/j.ijpsycho.2013.05.007. Epub 2013 May 18. PMID 23688673
- [Background] Taylor AE, Saint-Cyr JA, Lang AE. Frontal lobe dysfunction in Parkinson's disease. The cortical focus of neostriatal outflow. Brain. 1986 Oct;109 ( Pt 5):845-83. doi: 10.1093/brain/109.5.845. PMID 3779372
- [Background] Lenka A, Jhunjhunwala KR, Saini J, Pal PK. Structural and functional neuroimaging in patients with Parkinson's disease and visual hallucinations: A critical review. Parkinsonism Relat Disord. 2015 Jul;21(7):683-91. doi: 10.1016/j.parkreldis.2015.04.005. Epub 2015 Apr 17. PMID 25920541
- [Background] Abe Y, Kachi T, Kato T, Arahata Y, Yamada T, Washimi Y, Iwai K, Ito K, Yanagisawa N, Sobue G. Occipital hypoperfusion in Parkinson's disease without dementia: correlation to impaired cortical visual processing. J Neurol Neurosurg Psychiatry. 2003 Apr;74(4):419-22. doi: 10.1136/jnnp.74.4.419. PMID 12640053